CLINICAL TRIAL: NCT01747733
Title: Assessment of Sedation During Endoscopy, a Prospective Validation Study
Brief Title: Assessment of Sedation During Endoscopy
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jarno Jokelainen, MD, Principal Investigator, Helsinki University Central Hospital
Other Study IDs: DNRO 336/13/03/02/2012
Record Dates: First submitted 2012-12-07; First posted 2012-12-12 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Sedation
Keywords: Endoscopy; ERCP; PCS; Sedation; Bispectral index
MeSH Terms: interventions — Consciousness Monitors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Endoscopy patients: Patients undergoing endoscopy in the endoscopy unit in HUCH (Helsinki University Central Hospital).
  Interventions: Device: Bispectral Index

INTERVENTIONS:
Device: Bispectral Index — use of BiS-monitor in the assessment of the level of sedation in patients receiving sedation in endoscopy procedures when compared to clinical sedation scales, such as the Richmond agitation-sedation score.

SUMMARY:
Use of sedation is often required in endoscopic procedures such as ERCP (endoscopic retrograde cholangiopancreatography). However, assessment of the level of sedation during these procedures is not investigated in detail.

The purpose of this study is to compare different sedation scales and bispectral index during sedation in endoscopic procedures in order to find the best suited assessment method for sedation under these conditions.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing endoscopic procedure in the endoscopy unit in HUCH

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing endoscopic procedures requiring anaesthesist administered sedation in the endoscopy unit in HUCH
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
level of sedation | 1 day
  Sedation measured by Bispectral Index (BiS) compared with RASS (Richmond Agitation-Sedation Score), MOAA/S (Modified Observer's Assessment of Alertness/Sedation) and Ramsay sedation score

CONTACTS AND LOCATIONS:
Overall Officials: Jarno Jokelainen', M.D., Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

REFERENCES:
- [Background] Mazanikov M, Udd M, Kylanpaa L, Lindstrom O, Aho P, Halttunen J, Farkkila M, Poyhia R. Patient-controlled sedation with propofol and remifentanil for ERCP: a randomized, controlled study. Gastrointest Endosc. 2011 Feb;73(2):260-6. doi: 10.1016/j.gie.2010.10.005. PMID 21295639